CLINICAL TRIAL: NCT07164482
Title: "An Intermediate Size Patient Population Expanded Access Protocol to Evaluate the Safety and Efficacy of Allogeneic HB-adMSCs for the Treatment of Patients With Traumatic or Nontraumatic Brain Injury"
Brief Title: Intermediate Size Patient Population Expanded Access Protocol to Evaluate HB-adMSCs for the Treatment of Patients With Traumatic or Nontraumatic Brain Injury
Status: Available | Type: Expanded Access
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Other Study IDs: HBBI01
Record Dates: First submitted 2025-08-29; First posted 2025-09-10 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Brain Injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: HB- adMSCs (Hope Biosciences adipose derived mesenchymal stem cells) — Participants will receive allogenic HB-adMSCs through intravenous infusion only, with a treatment duration of 16 weeks, infusion rate 4-5mL/min and total volume of 250 mL Sodium chloride 0.9%. Each participant will receive a total of 6 doses of HB-adMSCs with a dosing regimen of approximately 2 weeks between infusion 1, infusion 2 and infusion 3, and 4 weeks between the remaining infusions.

SUMMARY:
This expanded access protocol is part of IND 031942 to evaluate efficacy and safety of multiple intravenous administrations of autologous HB-adMSCs for the treatment of nontraumatic or traumatic brain injury for up to 7 patients who passed pre-screening, completed screening, and were not randomized into the treatment group for the HBBI01 clinical study protocol entitled, "An Intermediate Size Patient Population Expanded Access Protocol to Evaluate the Safety and Efficacy of Allogeneic HB-adMSCs for the Treatment of Patients with Traumatic or Nontraumatic Brain Injury." under IND 027396.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 14 - 78 years of age
2. Patient should provide evidence of TBI or non -TBI as evidenced by documentation in their medical records and imaging that was done within the past 3 years.
3. Female participants of childbearing potential should not be pregnant or plan to become pregnant during protocol participation and for 6 months after the last investigational product administration. Female participants of childbearing potential should confirm the use of one of the following contraceptive measures:

   * Hormonal contraceptives associated with ovulation inhibition (oral, injectable, implantable, patch, or intravaginal).
   * Intrauterine device (IUD), or intrauterine hormone-releasing system (IUS).
   * Barrier contraceptive methods (condoms, diaphragm, etc.).
   * Surgery (occlusion bilateral tubal ligation, hysterectomy, vasectomized partner).

   OR

   Male participants if their sexual partners can become pregnant should ensure the use one of the following methods of contraception during protocol participation and for 6 months after the last administration of the investigated product:
   * Hormonal contraceptives associated with ovulation inhibition (oral, injectable, implantable, patch, or intravaginal).
   * Intrauterine device (IUD), or intrauterine hormone-releasing system (IUS).
   * Barrier contraceptive methods (condoms, diaphragm, etc.).
   * Surgery (vasectomy, occlusion bilateral tubal ligation (partner), hysterectomy (partner)).
4. Patient/LAR should be able to read, understand, and to provide voluntary consent.

Exclusion Criteria:

1. Women who are currently pregnant or lactating.
2. The patient has any active infection requiring medications per PI's discretion.
3. The patient has any clinical signs or symptoms of infection per PI's discretion.
4. The patient has hyperthermia or hypothermia.
5. The patient has any known recent (within the last 6 months) coagulation anomalies that are not being medically treated and are not stable per PI's discretion.
6. The patient has any abnormal laboratory values at the screening visit which the Investigator determines to be clinically significant and make the patient unsuitable for participation.
7. The Investigator determines the patient to be unsuitable for participation for other reasons, such as, but not limited to deep vein thrombosis (DVT), pulmonary embolus, cardiac arrhythmia, or those who have a prothrombotic condition, or who require persistent oxygen supplementation.

Ages: 14 Years to 78 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Hope Biosciences Research Foundation, Houston, Texas, United States